CLINICAL TRIAL: NCT05891613
Title: Liposomal Bupivacaine Versus 0.25% Bupivacaine Hydrochloride for Postoperative Analgesia After Breast Reduction Surgery: A Prospective, Single Blind, Non-randomized Controlled Trial
Brief Title: A Study of Liposomal Bupivacaine Versus 0.25% Bupivacaine Hydrochloride Post Breast Reduction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Basel A. Sharaf, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21-007358
Record Dates: First submitted 2023-05-26; First posted 2023-06-07 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Breast Reduction
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Breast Treatment Group: Bupivacaine Hydrochloride (Active Comparator): Subjects undergoing breast reduction surgery will receive standard 0.25% Bupivacaine Hydrochloride in one breast.
  Interventions: Drug: Bupivacaine Hydrochloride
- Treatment Breast Treatment Group: Liposomal (Exparel) Bupivacaine (Experimental): Subjects undergoing breast reduction surgery will receive a mixture of liposomal (Exparel) bupivacaine with plain 0.25% bupivacaine hydrochloride in contralateral breast.
  Interventions: Drug: Bupivacaine Hydrochloride; Drug: Liposomal Bupivacaine

INTERVENTIONS:
Drug: Bupivacaine Hydrochloride — 20 ml of 0.25% Bupivacaine (50 mg) with 20 ml of injectable saline (total of 40 cc) as a subcutaneous infiltration along the inframammary fold incision on one breast
Drug: Liposomal Bupivacaine — 20 ml of Liposomal (Exparel) Bupivacaine (266 mg/20 ml) on the contralateral breast
  Other Names: Exparel
  Arms: Treatment Breast Treatment Group: Liposomal (Exparel) Bupivacaine

SUMMARY:
The purpose of this research is to assess pain scores and opioid use when using Liposomal (Exparel) Bupivacaine versus Bupivacaine Hydrochloride.

DETAILED DESCRIPTION:
This is a prospective, multi-surgeon, single blind, non-randomized, controlled trial with breasts allocated to two parallel groups: A mixture of liposomal (Exparel) bupivacaine with plain 0.25% bupivacaine hydrochloride will be used on one side (Treatment side) as local infiltration, and plain 0.25% Bupivacaine Hydrochloride will be used in the control arm. Each breast will serve as the control for the other. The study is designed to evaluate early postoperative pain control of each of the products up to 72 hours postoperatively. These treatments are standard of care in clinical practice.

ELIGIBILITY:
Inclusion Criteria

- Adult female patients (18-70 years old) with symptomatic macromastia scheduled for breast reduction using a Wise pattern incision design.

Exclusion Criteria

* Inability to provide informed consent
* Medical or surgical history precluding breast reduction
* History of significant chronic pain requiring daily use of opioid or nonopioid analgesics
* Pregnancy
* Concomitant non-breast surgical procedure
* Previous chest wall irradiation
* Previous breast implant, breast reduction or breast lift surgery
* Known allergy to bupivacaine or liposomal bupivacaine
* Liver or kidney dysfunction
* Use of antiplatelet or anticoagulation therapy.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2024-01-24 (Actual); Primary Completion 2025-10-06 (Actual); Study Completion 2025-10-06 (Actual)

PRIMARY OUTCOMES:
Pain Scores in the first 72 hours post-operatively following breast reduction | 72 hours post-operatively
  Measured using validated self-reported Numerical Pain Rating Scale (NPRS). Participants rate pain using a scale of 0=none and 10=most severe.

CONTACTS AND LOCATIONS:
Overall Officials: Basel Sharaf, MD, DDS, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Minnesota, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No